CLINICAL TRIAL: NCT01213082
Title: Phase I/II Prospective, Randomized, Double-blinded Study of Intravitreal Anti-VEGF Therapy Combined With Proton Beam Radiation Versus Sham Irradiation in Treating Exudative Age-related Macular Degeneration
Brief Title: ProspectiveTrial of Proton Beam Combined With Anti-VEGF Therapy for Exudative Age-related Macular Degeneration (AMD)
Acronym: PBAMD2
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of California, Davis (Other)
Collaborators: University of California, San Francisco (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 223071
Record Dates: First submitted 2010-09-29; First posted 2010-10-01 (Estimated); Results first posted 2018-07-17 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-05

CONDITIONS: Exudative Age-related Macular Degeneration
Keywords: Exudative Age-related Macular Degeneration; Proton beam irradiation; ranibizumab; bevacizumab; anti-VEGF therapy

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- 24GyE + anti-VEGF (Experimental)
  Interventions: Drug: 24GyE proton and Anti-VEGF
- 16GyE + anti-VEGF (Experimental)
  Interventions: Drug: 16GyE and anti-VEGF
- Sham Irradiation + anti-VEGF (Sham Comparator)
  Interventions: Drug: Sham Irradiation and anti-VEGF

INTERVENTIONS:
Drug: 24GyE proton and Anti-VEGF — 24GyE proton beam will be administered in 2 fractions 24 hrs apart 2 to 6 weeks after intravitreal anti-VEGF therapy
  Other Names: 24Gy Proton Beam + Anti-VEGF
  Arms: 24GyE + anti-VEGF
Drug: 16GyE and anti-VEGF — 16GyE of Proton Beam Irradiation will be administered in 2 fractions 24 hrs apart 2 to 6 weeks after intravitreal anti-VEGF therapy
  Other Names: 16Gy proton beam + Anti-VEGF
  Arms: 16GyE + anti-VEGF
Drug: Sham Irradiation and anti-VEGF — 2 Sessions of Sham Proton Beam Irradiation 24 hrs apart administered 2 to 6 weeks after intravitreal anti-VEGF therapy
  Other Names: Sham proton beam + anti-VEGF
  Arms: Sham Irradiation + anti-VEGF

SUMMARY:
The purpose of this study is to test the hypothesis that proton beam irradiation combined with intravitreal anti-VEGF therapy is safe and potentially more effective than intravitreal anti-VEGF therapy alone in eyes with exudative age-related macular degeneration.

DETAILED DESCRIPTION:
Radiation combined with anti-VEGF therapy has been shown to be synergistic in treating cancer and result in sustained tumor regression. On-going clinical trials have shown potential synergism between intravitreal anti-VEGF therapy and epiretinal brachytherapy administered during vitrectomy surgery in treating eyes with exudative age-related macular degeneration (eAMD). In this study, we test the hypothesis that radiation to the macula administered noninvasively via proton beam is well-tolerated in eyes with eAMD when combined with intravitreal anti-VEGF therapy and that this combination therapy may act synergistically to result in sustained treatment effect in eyes with eAMD.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be eligible if the following criteria are met:

  * Ability to provide written informed consent and comply with study assessments for the full duration of the study
  * Age > 50 years
  * Patient related considerations
  * Able to maintain follow-up for at least 24 months.
  * Women must be postmenopausal without a period for at least one year.
  * Diagnosed with Age-related Macular Degeneration (ARMD) with active subfoveal choroidal neovascular membrane (CNVM), newly diagnosed or treated with first dose of anti-VEGF therapy within 6 weeks of enrollment
  * Visual acuity 20/40 to 20/400
  * Lesion size < 12 Disc Area
  * Submacular hemorrhage less than 75% of total lesion and not involving foveal center
  * Submacular fibrosis less than 25% of total lesion
  * Candidate for intravitreal anti-VEGF therapy

Exclusion Criteria:

* Subjects who meet any of the following criteria will be excluded from this study:

  * Prior enrollment in the study
  * Pregnancy (positive pregnancy test) or lactation
  * Any other condition that the investigator believes would pose a significant hazard to the subject if the investigational therapy were initiated
  * Participation in another simultaneous medical investigation or trial
  * Previous treatment with Photodynamic Therapy (PDT) or thermal laser in study eye
  * Anti-VEGF therapy within 6 weeks
  * Intravitreal or subtenon's Kenalog within 6 months
  * Intraocular surgery within 3 months or expected in the next 6 months
  * Current or planned participation in other experimental treatments for wet AMD
  * Other concurrent retinopathy or optic neuropathy
  * Other causes of CNVM, i.e. myopic degeneration or ocular histoplasmosis (POHS)
  * Significant media opacity precluding adequate view of the fundus for exam, photography or OCT
  * History of radiation therapy to the head or study eye
  * Diabetes mellitus or hemoglobin A1c > 6
  * Head tremor or h/o claustrophobia precluding positioning for proton irradiation
  * Inability to maintain steady fixation with either eye
  * History of Malignancy treated within 5 years
  * Allergy to Fluorescein dye

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2010-09; Primary Completion 2017-01-31 (Actual); Study Completion 2017-01-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Susanna S Park, MD PhD, Principal Investigator — University of California, Davis
Locations (1):
- University of California Davis Eye Center, Sacramento, California, United States

REFERENCES:
- [Derived] Evans JR, Igwe C, Jackson TL, Chong V. Radiotherapy for neovascular age-related macular degeneration. Cochrane Database Syst Rev. 2020 Aug 26;8(8):CD004004. doi: 10.1002/14651858.CD004004.pub4. PMID 32844399

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | 24GyE + Anti-VEGF | 16GyE + Anti-VEGF | Sham Irradiation + Anti-VEGF
Started | 12 | 11 | 11
Completed | 6 | 4 | 6
Not Completed | 6 | 7 | 5
Not completed — Lost to Follow-up | 6 | 7 | 4
Not completed — Physician Decision | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | 24GyE + Anti-VEGF | 16GyE + Anti-VEGF | Sham Irradiation + Anti-VEGF | Total
Number analyzed (Participants) | 12 | 11 | 11 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0 | 0
  Between 18 and 65 years | 0 | 0 | 0 | 0
  >=65 years | 12 | 11 | 11 | 34
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 6 | 6 | 6 | 18
  Male | 6 | 5 | 5 | 16
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 0 | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 0 | 0
  White | 12 | 11 | 11 | 34
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 12 | 11 | 11 | 34
best corrected visual acuity [Mean (Standard Deviation); unit: logMAR BCVA] | 0.72 (0.39) | 0.59 (0.51) | 0.55 (0.18) | 0.62 (0.38)

OUTCOME MEASURES:

1. Primary Outcome: Percent of Eyes With Severe Ocular Adverse
Description: vision loss of 3 or more lines associated with radiation retinopathy or papillopathy
Time Frame: Month 24
Measure: Number; unit: percentage of participants
Groups:
- 24GyE PBT: intravitreal anti-VEGF combined with 24GyE PBT for exudative AMD
- 16GyE PBT: intravitreal anti-VEGF combined with 16GyE PBT for exudative AMD
- Sham Radiation: intravitreal anti-VEGF combined with sham PBT for exudative AMD
Arm/Group | 24GyE PBT | 16GyE PBT | Sham Radiation
Number analyzed (Participants) | 6 | 4 | 6
percentage of participants | 0 | 0 | 0

2. Secondary Outcome: Number of Anti-VEGF Injections Administered
Description: efficacy measure
Time Frame: Month 24
Measure: Mean (Standard Deviation); unit: number of anti-VEGF injections per eye
Arm/Group | 24GyE PBT | 16GyE PBT | Sham Radiation
Number analyzed (Participants) | 6 | 4 | 6
number of anti-VEGF injections per eye | 4.67 (1.9) | 7.25 (2.1) | 9.67 (3.5)

ADVERSE EVENTS:
Time Frame: 24 months
Arm/Group | 24GyE + Anti-VEGF | 16GyE + Anti-VEGF | Sham Irradiation + Anti-VEGF
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/4 | 0/6
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/4 | 0/6
Other Adverse Events (participants affected / at risk) | 0/6 | 1/4 | 2/6
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | 24GyE + Anti-VEGF (N=6) | 16GyE + Anti-VEGF (N=4) | Sham Irradiation + Anti-VEGF (N=6)
Mild retinal vasculopathy possible radiation retinopathy (Eye disorders) | 0 (0) | 1 (1) | 2 (2) — as accessed at month 24
cataract progression due to radiation (Eye disorders) | 0 (0) | 0 (0) | 0 (0) — as assessed at month 24

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2010-09-08): https://cdn.clinicaltrials.gov/large-docs/82/NCT01213082/Prot_SAP_000.pdf